CLINICAL TRIAL: NCT05631067
Title: Feasibility and Acceptability of Remote Blood Pressure Monitoring and Risk Stratification in the Fourth Trimester to Reduce Maternal Cardiovascular Morbidity and Mortality in Nigeria
Brief Title: Feasibility and Acceptability of Risk Stratification in the Fourth Trimester to Reduce Maternal Morbidity and Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Abuja Teaching Hospital (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud, Instructor of Medicine (Principal Investigator), Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #202207009
Record Dates: First submitted 2022-09-14; First posted 2022-11-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP monitoring arm (Experimental): Participants will be adults >18 years of age admitted for delivery with a diagnosis of HDP (i.e., chronic hypertension, gestational hypertension, preeclampsia, eclampsia, the HELLP syndrome, or chronic hypertension with superimposed preeclampsia) per the American College of Obstetricians and Gynecologists Criteria.
  Interventions: Behavioral: Remote blood pressure monitoring; Diagnostic Test: NT proBNP assessment
- Control arm (Active Comparator): Control participants will be adults >18 years of age with an uncomplicated pregnancy and delivery, and without a diagnosis of HDP.
  Interventions: Diagnostic Test: NT proBNP assessment

INTERVENTIONS:
Behavioral: Remote blood pressure monitoring — Participants will receive a blood pressure monitor to check daily BPs for two weeks post partum
  Arms: BP monitoring arm
Diagnostic Test: NT proBNP assessment — Participants will have biomarker assessment at 0-2 days postpartum

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are major causes of maternal morbidity and mortality globally and are associated with peripartum and future cardiovascular disease, including stroke, heart failure, and myocardial infarction. About 1 out of every 10 maternal deaths in Sub-Saharan Africa are associated with HDP, and most of these deaths are preventable with timely, implementation of evidence-based strategies, including postpartum blood pressure (BP) monitoring, treatment of elevated BP and comprehensive postpartum follow up as recommended by the American College of Obstetricians and Gynecologists (ACOG) and the World Health Organization (WHO).

This study aims to contextualize, implement, and evaluate the feasibility, fidelity, and acceptability of: 1) postpartum remote blood pressure monitoring and 2) NTproBNP testing for postpartum risk stratification in women with HDP at the University of Abuja Teaching Hospital in the Federal Capital Territory of Nigeria

DETAILED DESCRIPTION:
Aims:

1. To evaluate the feasibility, fidelity, and acceptability of home blood pressure monitoring in postpartum patients (n=90) with HDP. The investigators hypothesize that remote blood pressure monitoring will be feasible, implemented as intended, and acceptable among patients, physicians, and other health care workers to improve awareness and early diagnosis of elevated blood pressures (>140/90 mm Hg) in postpartum patients with HDP.
2. To evaluate the association between N Terminal-proBNP (NT-proBNP) levels and short-term cardiovascular outcomes (i.e., all-cause cardiovascular hospital readmission, postpartum pre-eclampsia, hypertensive urgency/emergency, stroke, heart failure/pulmonary edema, seizure and mortality at 12-weeks postpartum) in patients with HDP.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Admitted for delivery
* Clinical diagnosis of HDP (i.e., chronic hypertension, gestational hypertension, preeclampsia, eclampsia, the HELLP syndrome, or chronic hypertension with superimposed preeclampsia)

Control participants:

* Adults >18 years of age
* Admitted for delivery
* with an uncomplicated pregnancy and delivery

Exclusion Criteria:

* Unable to provide consent
* Unable to check blood pressure at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | Through study completion at 1 year
  Number of participants recruited

SECONDARY OUTCOMES:
Fidelity | 2 weeks
  10 daily home BP checks per participant during 2-week study period
Retention | 2 weeks
  Proportion (95% CI) of participants who remained with the home BP monitoring pilot study for the 14-day period

OTHER OUTCOMES:
Exploratory Outcome | 2 weeks
  Detection of elevated BP>140/90 mm Hg
  Detection of elevated BP>140/90 mm Hg
Incidence of combined adverse cardiovascular events | 12 weeks
  The incidence of a combined adverse cardiovascular endpoint (all-cause cardiovascular hospital readmission, postpartum pre-eclampsia, hypertensive urgency/emergency, stroke, heart failure/pulmonary edema, seizure and mortality) at 12-weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Mahmoud, MD, Principal Investigator — Washington University School of Medicine; Mark D Huffman, MD MPH, Principal Investigator — Washington University School of Medicine; Dike Ojji, MBBS PhD, Principal Investigator — University of Abuja Teaching Hospital; Kathryn Lindley, MD, Principal Investigator — Vanderbilt University
Locations (1):
- University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available within 1 year of study completion
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion
Access Criteria: Criteria and URL will be provided